CLINICAL TRIAL: NCT00524108
Title: Retrospective Analysis of Clinical Features in Ventriculoperitoneal Shunt Infections and Time to Re-Implantation in Adults
Brief Title: Retrospective Analysis of Clinical Features in Ventriculoperitoneal Shunt Infectionsin Adults
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: PRO07080212
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Ventriculoperitoneal Shunt; Infection
Keywords: shunt; internal ventriculoperitoneal
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objectives of this study are:

* To describe the incidence of clinical features in adults with internal ventriculoperitoneal (VP) shunt infections,
* To determine the validity of laboratory parameters in adults with internal ventriculoperitoneal shunt infections and
* To evaluate the relationship between the timing of shunt re-implantation with the rates of relapse and secondary infection.

DETAILED DESCRIPTION:
Information from medical records of patients seen by the PI will be collected and analyzed to describe the incidence of clinical features in adults with internal ventriculoperitoneal shunt infections, to determine the validity of laboratory parameters in adults with internal ventriculoperitoneal shunt infections and to evaluate the relationship between the timing of shunt re-implantation with the rates of relapse and secondary infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age >= 18 yrs) with VP shunts (ventriculoatrial [VA], and other cerebrospinal fluid [CSF] catheters will not be included).
* Cases will include patients with a diagnosis of VP shunt infection.
* Controls will be patients with a clinical suspicion of shunt infections with negative CSF cultures.

Exclusion Criteria:

* Patients with meningitis from community acquired organisms (e.g. Streptococcus pneumoniae, Neisseria meningitidis, Listeria monocytogenes and Haemophilus Influenzae).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: VP shunt infection
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adarsh Bhimraj, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States